CLINICAL TRIAL: NCT06899438
Title: Does Botulinum Toxin Type-A an Effective Way of Relieving Pain in Myofascial Pain Syndrome or Not
Brief Title: Does Botulinum Toxin Type-A Injection an Effective Way of Relieving Pain in Myofascial Pain Syndrome Patients or Not
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Taner Dandinoğlu, Principal investigator, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-PMR-1
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Myofacial Pain Syndromes
Keywords: Myofascial pain; Botulinum toxin; Prilocaine; İnjection
MeSH Terms: conditions — Facial Neuralgia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botulinum toxin injection group (BIG) (Experimental)
  Interventions: Drug: Botulinum Toxin A Injection
- Prilocaine injection group (PIG) (Active Comparator)
  Interventions: Drug: Prilocaine HCl % 2 injectable solution

INTERVENTIONS:
Drug: Botulinum Toxin A Injection
  Arms: Botulinum toxin injection group (BIG)
Drug: Prilocaine HCl % 2 injectable solution
  Arms: Prilocaine injection group (PIG)

SUMMARY:
In this research prilocaine and botulinum toxin (BoNT-A) interventions prospectively compared to find out the effect of BoNT-A injection on myofascial pain syndrome (MPS).

The main question it aims to answer is: Does Botulinum Toxin Type-A an Effective Way of Relieving Pain in Myofascial Pain Syndrome or not?

For this purpose thirty-eight patients randomly assigned into two study groups. While BoNT-A injection group (BIG group n=19) treated with 20 units of toxin to each trigger point (TP), remaining treated with 2 ml prilocaine (PIG group n=19) with same procedure.

Pre-treatment, 2nd and 6th weeks findings were clinically recorded.

DETAILED DESCRIPTION:
Visual Analog Scale (VAS), 4-Point Verbal Rating Scale (VRS), Pain Pressure Threshold (PPT), Short Form-36 (SF-36) and Beck Depression Inventory (BDI) tools were used to evaluate findings of the research.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 20 years

Presence of myofascial pain syndrome (MPS) symptoms for more than 3 months

Ability and willingness to provide written informed consent

Exclusion Criteria:

Any injection to trigger points within the last 2 months

Diagnosis of fibromyalgia syndrome

Presence of significant respiratory or cardiovascular disease

Presence of psychiatric disorders that may interfere with study participation

History of shoulder or cervical spine intervention within the last year

Presence of cervical myelopathy or cervical radiculopathy

Inability to cooperate with study procedures or assessments

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2009-08-26 (Actual); Primary Completion 2010-01-26 (Actual); Study Completion 2010-01-26 (Actual)

PRIMARY OUTCOMES:
Visual analog scale, 4-point verbal rating scale, Pressure pain threshold | Pre-treatment, 2nd and 6th week scores were recorded.
  Visual analog scale (VAS) between 0 and 10 was used to measure subjective complaints of pain (0 painless-10 worst pain).
  4-point verbal rating scale (VRS) was also used to evaluate the affected area covering the TP (3 Severe pain; strong verbal response, accompanied by grimacing of face, withdrawal of hand, 2 Modarate pain, complaint reported spontaneously or mostly response to asking, accompanied by behavioral changes like grimacing, 1 Mild pain, pain is expressed when questioning without behavioral responces and 0 None, no pain).
  An algometry device is used to evaluate "Pressure pain threshold" (PPT) and the sensitivity that the person felt is recorded in kg.

CONTACTS AND LOCATIONS:
Overall Officials: Baki Özdemir, MD, Principal Investigator — LHU Ankara Hospital Department of Rheumatology

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study are available from Military Medical Academy of Turkish Army but restrictions apply to the availability of these data (All patients are retired or active soldiers and their spouses) and so are not publicly available. However, under appropriate circumstances findings are available from the author upon reasonable request. If it is requested, data will be available for reviewers from Dr Taner Dandinoglu, E-mail: dandinoglu@gmail.com.

REFERENCES:
- Available data/document: Clinical Study Report — https://tez.yok.gov.tr/UlusalTezMerkezi/tezDetay.jsp?id=ojJkM_gxQRaH4Sn9fMdQWw&no=8WIZbpBlZOGWvkUUwksxFg